CLINICAL TRIAL: NCT01357213
Title: A Phase I, Blinded, Placebo-controlled, Dose-escalation Study of the Safety and Pharmacokinetics of XOMA 3AB Administered Intravenously in Healthy Adults
Brief Title: Phase 1 PK Study of XOMA 3AB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-0091; N01AI80026C
Record Dates: First submitted 2011-05-05; First posted 2011-05-20 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2013-05

CONDITIONS: Botulism
Keywords: Botulism, Clostridium
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Arm 2 (Placebo Comparator): Placebo in all three cohorts
  Interventions: Other: Placebo
- Arm 1 (Experimental): XOMA 3AB in 3 dose levels/cohorts A, B or C.
  Interventions: Drug: XOMA 3AB

INTERVENTIONS:
Drug: XOMA 3AB — Single intravenous infusion of XOMA 3AB in three cohorts at different concentrations.
  Arms: Arm 1
Other: Placebo — Normal saline 100 ml
  Arms: Arm 2

SUMMARY:
This is a phase I, single-center, placebo-controlled, double-blinded, dose escalation study of anti-botulinum toxin monoclonal antibodies in healthy adult volunteers. Volunteers will be hospitalized in the Johns Hopkins Phase 1 unit during the infusion and until after the 24-hour blood draw. Three escalating dose cohorts of a combination of three anti-botulinum monoclonal antibodies will be evaluated. Each cohort will consist of eight volunteers in which they will receive a single intravenous infusion of active drug or placebo. Placebo will be normal saline. Volunteers will be followed for safety for up to 120 days after infusion depending on dose cohort.

DETAILED DESCRIPTION:
This is a phase I, single-center, placebo-controlled, double-blinded, dose escalation study of anti-botulinum toxin monoclonal antibodies in healthy adult volunteers. Volunteers will be hospitalized in the Johns Hopkins Phase 1 unit during the infusion and until after the 24-hour blood draw. Three escalating dose cohorts of a combination of three anti-botulinum monoclonal antibodies will be evaluated. Each cohort will consist of eight volunteers in which they will receive a single intravenous infusion of active drug or placebo. Placebo will be normal saline. Volunteers will be followed for safety for up to 120 days after infusion depending on dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent understood and signed
* Healthy male or healthy, non-pregnant, non-lactating female
* Willingness to comply and be available for all protocol procedures
* Age between 18 and 45 years, inclusive on the day of infusion
* Body Mass Index of < 35
* Blood pressure within acceptable limits (systolic blood pressure </=140mmHg and diastolic blood pressure </=90mmHg). If subject is receiving anti-hypertensive medications, blood pressure must be well controlled with no changes in anti-hypertensive medications for at least 3 months.
* If the subject is female and of childbearing potential, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to infusion.
* If the subject is female and of childbearing potential, she agrees to practice abstinence from sexual intercourse with men or use acceptable contraception, for the duration of the study:

  * A woman is considered of childbearing potential unless post-menopausal (>/= 1 year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)
  * Acceptable contraception methods are restricted to effective devices (Intrauterine Contraceptive Devices (IUDs), NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, condoms with spermicidal agents, monogamous relationship with a vasectomized partner, or successful Essure placement with documented confirmation test at least 3 months after the procedure.
* All requested screening laboratory values are within the range specified in the table, "Acceptable Ranges of Screening Labs and Vital Sign Measurements" (Appendix B).
* Has adequate venous access for the infusion.
* The drug screen is negative
* Breathalyzer test is negative.

Exclusion Criteria:

* History of a chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart or nervous system, or other metabolic and autoimmune/inflammatory conditions that would either interfere with the accurate assessment of the objectives of the study or increase the risk profile of the subject such as:

  * Diabetes
  * Asthma requiring use of medication in the year before screening
  * Autoimmune disorder, such as lupus, Wegener's, rheumatoid arthritis
  * Coronary artery disease
  * History of malignancy except low-grade (squamous and basal cell) skin cancer thought to be cured
  * Chronic renal hepatic or pulmonary disease (except previous asthma which has required no treatment for the past year)
  * History of severe allergic reaction of any type to medications, bee stings, food, or environmental factors or hypersensitivity or reaction to immunoglobulins. Severe allergic reaction is defined as any of the following:

    * Anaphylaxis
    * Urticaria
    * Angioedema
  * A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds)
  * Clinically significant abnormal electrocardiogram at screening in the judgment of the investigator
* Positive serology results for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (HBsAg), or Hepatitis C Virus (HCV) antibodies
* Febrile illness with temperature >37.6°C within 7 days of dosing
* Pregnant or breastfeeding
* Donated blood within 56 days of enrollment
* Known allergic reactions to any of the study product components present in the formulation or in the processing, as listed in the Investigator Brochure.
* Treatment with another investigational drug within 30 days of dosing
* Receipt of a monoclonal antibody at any time in the past
* Receipt of antibody (e.g. TIG, VZIG, IVIG, IM gamma globulin) or blood transfusion within 6 months or within 5 half-lives of the specific product given
* Receipt of any live vaccines within the previous 3 months or within 5 half-lives of the specific vaccine given
* Receipt of any killed vaccines within the previous 1 month
* Lack of ability to fully understand the informed consent (e.g. cannot speak or read English)
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Use of H1 antihistamines or beta-blockers within 5 days of dosing.
* Use of any of the following medications within 30 days prior to study entry or planned use during the study period:

  * immunosuppressives (except Nonsteroidal Anti-Inflammatory Drugs (NSAIDS))
  * immune modulators
  * oral corticosteroids (topical steroids are acceptable)
  * anti-neoplastic agents
  * any vaccine (licensed or investigational)
* Previous exposure to botulinum toxin, receipt of antibodies against botulinum toxin, or previous treatment with equine antitoxin
* Any previous injection or planned injection within 12 months after enrollment of botulinum toxin for cosmetic reasons, spastic dysphonia, torticollis, or any other reason
* Any specific condition that in the judgment of the investigator precludes participation because it could affect subject safety;
* Co-enrollment in another study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of XOMA 3AB: occurrence of adverse events and serious adverse events. | Day 0 to Day 90 and to Day 120 (depending on dose cohort).
Safety and tolerability of XOMA 3AB: Changes from baseline in vital signs, physical examinations, chemistry and complete blood count with differential laboratory studies, dipstick urinalysis, and electrocardiograms. | Day 0, 1, 2, 3, 7, 14, 28, 42, 56, Day 90 and to 120 days (depending on dose cohort).

SECONDARY OUTCOMES:
Immunogenicity: measuring Human anti-human antibodies (HAHA) to XOMA 3AB | Day 0, 28, 56, 90 and 120 days (depending on dose cohort).
Pharmacokinetics of XOMA 3AB:Area under the curve to the last time with a measurable value (AUC(0-t)) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Volume of distribution (Vz) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Total clearance (CL) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Elimination half-life (t½) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Elimination rate constant (gimel z) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Area under the curve to infinity (AUC(inf)) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Time to Cmax (Tmax) measured from end of infusion | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Maximum plasma titer/concentration (Cmax) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)
Pharmacokinetics of XOMA 3AB: Mean residence time (MRT) | Serially on day 0, 1, 2, 3, 7, 14, 28, 42, 56, 90 and 120 days (depending on dose cohort)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland, United States

REFERENCES:
- [Background] Nayak SU, Griffiss JM, McKenzie R, Fuchs EJ, Jurao RA, An AT, Ahene A, Tomic M, Hendrix CW, Zenilman JM. Safety and pharmacokinetics of XOMA 3AB, a novel mixture of three monoclonal antibodies against botulinum toxin A. Antimicrob Agents Chemother. 2014 Sep;58(9):5047-53. doi: 10.1128/AAC.02830-14. Epub 2014 Jun 9. PMID 24913160